CLINICAL TRIAL: NCT02739243
Title: Addressing the Hidden Patient - A Randomised-controlled Trial of a Tailored Group Intervention for Caregivers of Cancer Patients (PREPARE)
Brief Title: A Clinical Trial on a Group Treatment for Distressed Caregivers of Cancer Patients
Acronym: PREPARE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrolment slower than anticipated accrual.
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Markus Haun, MD, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-655/2015; ISRCTN22231701 (Registry Identifier: ISRCTN registry)
Record Dates: First submitted 2016-04-07; First posted 2016-04-15 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Distress in Caregivers of Cancer Patients

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored group intervention (Experimental): Participants take part in the tailored group intervention which consists of five 90-minute group sessions over eight weeks. The sessions are in the form of structured group talk/discussions following specific themes:
  Session 1 - Coping and acceptance: identification of common themes from participants' feedback, provision of information about support services, mindfulness practices
  Session 2 - Distress: introduction of the distress model, identification of resources, breathing practices
  Session 3 - Handling of stressful situations: individual identification in tandems, discussion of common pitfalls in the group
  Session 4 - Self-care: inspection of individual daily routines, group collects positive experiences with "windows" for self-care
  Session 5 - Feedback and outlook: stabilisation, retrospective reflection on the group experience and its benefits and, if applicable, potential adverse events
  Interventions: Behavioral: Tailored group intervention (PREPARE)
- Treatment as usual (Active Comparator): Participants are provided with brief information in a leaflet, about the possibilities for individual counselling including referral to the local outpatient cancer counselling centre providing client-centred counselling and financial social work.
  Interventions: Behavioral: Individual treatment as usual

INTERVENTIONS:
Behavioral: Tailored group intervention (PREPARE)
  Arms: Tailored group intervention
Behavioral: Individual treatment as usual
  Arms: Treatment as usual

SUMMARY:
Background and study aims: Being a caregiver for someone with cancer can be very difficult emotionally. For many the patient is a family member or friend, and so this can cause the caregiver a great deal of psychological distress. There are currently very few studies looking into the effectiveness of psychological treatments for distressed caregivers of cancer patients. This study is looking at tailored group therapy program for carers of cancer givers. The aim of this study is to find out whether this program can help to lower levels of distress in cancer caregivers and help them to better cope with caring for someone with the illness.

ELIGIBILITY:
Inclusion Criteria:

1. Time since initial diagnosis (of patient) not longer than six months previously
2. Significant distress against the background of the cancer disease (QSC-R10C exceeding 16 points)
3. Provision of informed consent
4. Aged 18 or over, either gender

Exclusion Criteria:

1. Inability to give informed consent
2. Insufficient German language knowledge
3. Cognitive impairment impeding handling of questionnaires
4. Severe psychiatric disease (acute psychosis or acute suicidality)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Distress | change from baseline distress at 1 week post treatment
  measured using the Questionnaire on Stress in Caregivers of Cancer Patients Revised version (QSC-R10C)

SECONDARY OUTCOMES:
Depression | change from baseline depression at 1 week post treatment and at 6 months post treatment
  measured using the Patient Health Questionnaire-9 (PHQ-9)
Anxiety | change from baseline anxiety at 1 week post treatment and at 6 months post treatment
  measured using the Generalized Anxiety Disorder-7 (GAD-7)
General distress | change from baseline general distress at 1 week post treatment and at 6 months post treatment
  measured using the Distress Thermometer (NCCN DT)
Unmet needs | change from baseline unmet needs at 1 week post treatment and at 6 months post treatment
  measured using the Supportive Care Needs Survey - Partners & Caregivers (SCNS-P&C-G)
Self-efficacy in coping with the cancer disease | change from baseline self-efficacy at 1 week post treatment and at 6 months post treatment
  measured using the adapted General Perceived Self-Efficacy Scale
Utilisation of primary healthcare | change from baseline to 1 week post treatment and 6 months post treatment
  measured via the number of visits with the individual primary care physician
Positive bonding with the group | change from baseline bonding at 1 week post treatment and 6 months post treatment
  measured via the Positive Bonding Scale of the Group Questionnaire (GQ-D)

CONTACTS AND LOCATIONS:
Overall Officials: Markus W Haun, MD, Principal Investigator — Department of General Internal Medicine and Psychosomatics, Heidelberg University Hospital

IPD SHARING:
Plan to Share IPD: Undecided